CLINICAL TRIAL: NCT00643513
Title: Quality Of Life And Symptoms In Postmenopausal Women With Hormone Receptor Positive Disseminated Breast Cancer While Receiving Faslodex.
Brief Title: Quality Of Life While Receiving Faslodex
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca Russia, Clinical Study Information
Other Study IDs: NIS-ORU-FAS-2007/1
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: QUALITY OF LIFE; POSTMENOPAUSAL WOMEN; HORMONE RECEPTOR POSITIVE DISSEMINATED BREAST CANCER; FASLODEX
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
To study QoL related response, symptom spectrum and severity in disseminated breast cancer patients receiving Faslodex hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic and/or cytological proven breast cancer.
* Patients with metastases of breast cancer ± postmenopausal primary tumor ≥12 months.
* Positive oestrogen receptors (ER+), positive progesterone receptors (PgR+) or unknown hormonal receptors (if duration between surgery and metastasis occurring is not less 2 years) which are indirect confirmation of hormone sensitive tumor.
* ECOG performance status of ≤ 2
* Patient willingness to take part in the programm
* Life expectancy of more than 6 months.
* Patient ability to complete a questionnaire.

Exclusion Criteria:

* Contraindications for Faslodex therapy
* Other anticancer therapy (chemotherapy, hormonal therapy with other drugs, radiotherapy), except for radiotherapy of sites which are not only measurable or evaluable manifestation of disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-06; Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To study QoL related response, symptom spectrum and severity in disseminated breast cancer patients receiving Faslodex hormonal therapy.

CONTACTS AND LOCATIONS:
Locations (24):
- Russia (24):
  - Research Site, ?rasnodar
  - Research Site, Astrakhan
  - Research Site, Blagoveshenk
  - Research Site, Chita
  - Research Site, Igevsk
  - Research Site, Kemerovo
  - Research Site, Kursk
  - Research Site, Magadan
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Penza
  - Research Site, Petropavlovsk
  - Research Site, Rostov
  - Research Site, Saint Petersburg
  - Research Site, Salekhard
  - Research Site, Samara
  - Research Site, Shahti
  - Research Site, Surgut
  - Research Site, Tiva
  - Research Site, Tomsk
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Volgodonsk
  - Research Site, Yakutsk